CLINICAL TRIAL: NCT02144961
Title: Observational Study to Compare Research-only Breast Ultrasound to Standard of Care Physical Exam for Identifying Tissue Necrosis in Post-mastectomy Patients Undergoing Planned Breast Reconstruction.
Brief Title: The Effects of Indocyanine Green Angiography (IGA) on Deep Inferior Epigastric Artery Perforator (DIEP) Flap Design and Post-Operative Fat Necrosis
Acronym: SPY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Skye Stewart, Project Manager, University of Washington
Other Study IDs: 45728-A
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; Deep Inferior Epigastric Artery Perforator (DIEP); Indocyanine Green Angiography (IGA); autologous tissue transfer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound: Breast ultrasound in female patients who are post-mastectomy pursuing autologous tissue breast reconstruction surgery.

SUMMARY:
The aim of this study is to prospectively evaluate the effect of intra-operative Indocyanine green angiography (IGA) on both flap design and rate of post-operative fat necrosis in patients undergoing autologous breast reconstruction utilizing the Deep Inferior Epigastric Artery Perforator (DIEP) flap.

DETAILED DESCRIPTION:
For many post-mastectomy cancer patients seeking breast reconstruction, microsurgical, autologous tissue transfer is a desirable alternative to more conventional, implant-based procedures. In general terms, this technique entails use of one's own tissue, transferred from a distant anatomic site, to recreate the absent breast. This tissue, usually a composite of skin and subcutaneous adipose tissue, is isolated along with its source artery and vein, and transferred to the chest wall where it is connected (anastomosed) to a local blood supply.

Though there have been many donor tissues (flaps) described for this purpose, abdominal tissue supplied by small, perforating blood vessels originating from the deep inferior epigastric artery, has become the microsurgical gold standard. This so-called DIEP flap provides abundant tissue that can be easily sculpted to fill most breast defects with minimal donor site morbidity. Like all microvascular, free tissue transfers, however, the DIEP flap is not without its potential complications. One potential complication that is most distressing to patients occurs when a portion of the subcutaneous adipose tissue transferred exceeds the available blood supply. This devascularized fat eventually undergoes necrosis that may not only complicate the interpretation of future mammograms, but may result in palpable, painful, and occasionally visible, irregularities within the transferred tissue. Though many techniques/interventions/technologies have been described to minimize the incidence of fat necrosis, its occurrence remains frustratingly unpredictable and relatively common, with published rates ranging between 6 and 17 %.

In theory, maximizing perfusion to composite tissue flaps should minimize the rate of fat necrosis. As such, many techniques have emerged in DIEP flap surgery intended to maximize perfusion. One common technique is the use of pre-operative, CT angiography (CTA) to identify the largest and most anatomically favorable perforating vessels to include in the composite tissue transferred. Though elegant in its simplicity, use of this technique has never been demonstrated to decrease the rate of fat necrosis in DIEP reconstructions. In recent years, however, another technology intended to intra-operatively evaluate tissue perfusion has emerged that may prove very beneficial in the realm of microvascular free tissue transfer- Indocyanine green angiography (IGA).

IGA refers to the peripheral venous injection of lyophilized indocyanine green, a contrast agent that fluoresces when excited by a laser of specific wavelength A charge-coupled camera, held above the tissue of interest, can then detect the stimulated fluorescence and project an image of "real-time" tissue perfusion that is proportional to emission intensity. The application of IGA technology in reconstructive plastic surgery, a discipline that relies largely on immediate and accurate assessment of tissue perfusion, has recently generated much discussion.

We believe that perforator selection in DIEP breast reconstructions, a process traditionally dictated at our institution by pre-operative CTA, may be heavily influenced by intra-operative IGA. We further hypothesize that use of intra-operative IGA in DIEP breast reconstructions may reduce the incidence of post-operative fat necrosis.

The aim of this study is to prospectively evaluate the effect of intra-operative Indocyanine Green Angiography (IGA) on both flap design and rate of post-operative fat necrosis in patients undergoing autologous breast reconstruction utilizing the Deep Inferior Epigastric Artery Perforator (DIEP) flap.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients at the University of Washington
2. Aged twenty-five to sixty-five years
3. Pursuing immediate or delayed, DIEP-based, autologous, microsurgical breast reconstruction at the University of Washington Medical Center

Exclusion Criteria:

1. Patients unsuitable for autologous, microsurgical breast reconstruction utilizing the DIEP flap - i.e. patients who have undergone prior extensive abdominal surgeries, have inadequate abdominal tissue bulk, who cannot comply with standardized post-operative restrictions / assessments or patients afflicted with a medical condition(s) precluding prolonged general anesthesia and surgery.
2. Patients who have a known allergy to contrast media will also be excluded from this study.
3. Patients unable to read and write in English will be excluded.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females pursuing breast reconstruction after having undergone mastectomy. In the overwhelming majority of cases, this procedure is indicated for breast cancer treatment. Eligible patients will have their breast reconstruction done at the University of Washington Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Rate of post-operative fat necrosis | 3-6 months post-operatively
  Prospectively evaluate the effect of intra-operative IGA on both DIEP flap design, and rate of post-operative DIEP fat necrosis as compared by physical exam and breast ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States